CLINICAL TRIAL: NCT06438952
Title: Efficacy and Duration of Pain Relief in Transforaminal and Lumbar Sympathetic Blocks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E.142568
Record Dates: First submitted 2024-05-20; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain; Lumbar Disc Herniation
Keywords: Transforaminal Steroid İnjection; Lumbar Sympathetic Blockade; Lumbar Disc Herniation; Neuropathic Pain Questionnaire; Numerical Rating Scale
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addition of lumbar sympathetic blockade to transforaminal steroid injection (Active Comparator): The patient will receive both transforaminal steroid injection and lumbar sympathetic blockade.
  Interventions: Procedure: Transforaminal steroid injection combined with lumbar sympathetic blockade
- Transforaminal steroid injection only (Placebo Comparator): The patient will only receive transforaminal steroid injection.
  Interventions: Procedure: Transforaminal steroid injection only

INTERVENTIONS:
Procedure: Transforaminal steroid injection combined with lumbar sympathetic blockade — Transforaminal steroid injection will be made with 2 mg dexamethason + 20 mg lidocaine + 5mg bupivacaine + 5 mcg fentanyl + 100mg magnesium under US-guidance Lumbar sympathetic blockade will be made with 5 ml 0.5% bupivacaine + 6 mg dexamethason + 10 ml NaCl
  Arms: Addition of lumbar sympathetic blockade to transforaminal steroid injection
Procedure: Transforaminal steroid injection only — Transforaminal steroid injection will be made with 2 mg dexamethason + 20 mg lidocaine + 5mg bupivacaine + 5 mcg fentanyl + 100mg magnesium under US-guidance
  Arms: Transforaminal steroid injection only

SUMMARY:
Low back pain is a symptom that is frequently seen in the general population and reduces the quality of life of patients. Conventional medical treatment for patients with low back pain includes oral medication, lifestyle modification, education, exercises, lumbar traction and manual manipulation, heat application, and other interventional procedures. Epidural injections, one of the interventional procedures, are one of the common treatment methods for low back pain, especially caused by disc prolapse. Steroids are commonly used to reduce inflammation in the epidural space. Epidural steroid injection can be given to the lumbar epidural space via transforaminal, interlaminar and caudal routes, and the effectiveness rate of each is different. These interventional methods used to treat low back pain can be applied in combination.

The main purpose of this study is to observe how adding lumbar sympathetic blockade will affect the patient's pain in the postoperative period in patients to whom we applied caudal epidural and transforaminal steroid injection.

DETAILED DESCRIPTION:
Low back pain is a symptom that is frequently seen in the general population and reduces the quality of life of patients. Conventional medical treatment for patients with low back pain includes oral medication, lifestyle modification, education, exercises, lumbar traction and manual manipulation, heat application, and other interventional procedures [1, 2]. Epidural injections, one of the interventional procedures, are one of the common treatment methods for low back pain, especially caused by disc prolapse. Steroids are widely used to reduce inflammation in the epidural space [3, 4]. Epidural steroid injection can be administered to the lumbar epidural space via transforaminal, interlaminar and caudal routes, and each has different efficacy rates [5-7].

Sympathetically maintained pain, including lumbar sympathetic ganglion block (LSGB), complex regional pain syndrome (CRPS) types I and II, neuropathies (such as postherpetic neuralgia, stump or phantom limb pain), diabetic polyneuropathy, and ischemic pain from vascular insufficiency in the lower leg It is a widely applied procedure for diagnosing and managing diseases [8]. The autonomic nervous system consists of sympathetic and parasympathetic departments. As the name suggests, blood supply to the lower extremity increases after lumbar sympathetic block. This is useful in sympathetic system-mediated treatment of pain [9].

The most important reason for adding fentanyl and magnesium as adjvams is to improve the quality of analgesia and provide analgesia for a longer period of time. Both fentanyl and magnesium have the ability to modulate neurotransmitter release and affect neuronal excitability. Fentanyl demonstrates the role of the sympathetic nervous system in modulating pain by increasing the effectiveness of endogenous opioids in the sympathetic ganglia and central nervous system. Magnesium competes with calcium; It reduces the release of neurotransmitters such as acetylcholine.

Magnesium's ability to inhibit the release of acetylcholine contributes to its anticonvulsant properties. Additionally, blocking NMDA receptors contributes to its analgesic effects. Additionally, magnesium's ability to enhance the effects of local anesthetics has been studied. By increasing the firing threshold in nerves and causing hyperpolarization, magnesium enhances the effect of local anesthetics, thereby improving nerve blockade. This enhancement of nerve blockade is particularly evident when magnesium is added to agents such as bupivacaine [10, 11].

These interventional methods used to treat low back pain can be applied in combination. There is not enough research on this subject.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III
* Patients who underwent facet joint injection and transforaminal injection due to lumbar disc herniation

Exclusion Criteria:

* Patients with known allergies to the drugs to be used in treatment
* Infection near the puncture site
* Known coagulation disorders
* Patients with internal fixation or severe anatomical variation such as scoliosis and tumor
* History of sympathetic chemical or thermal neurolysis
* Alcohol and drug use
* Disorder of consciousness
* Liver failure, renal failure, advanced cardiac failure
* Uncontrolled diabetes mellitus
* Morbid obesity (body mass index (BMI) > 35 kg m-2)
* Female patients during pregnancy and breastfeeding
* Not approving the informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity score | Preoperative and postoperative 24th hour, 1st week, 1st month and 6th month
  Postoperative pain assessed with numeric rating scale (NRS 0: no pain 10:pain as bad as can be )

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Preoperative and postoperative 24th hour, 1st week, 1st month and 6th month
Neuropathic pain questionnaire | Preoperative and postoperative 24th hour, 1st week, 1st month and 6th month
Patient satisfaction | Patient satisfaction measured using a numeric rating scale 0 to 10 (0 = unsatisfied; 10 =very satisfied)
  The patient is asked to give a score between 1 and 10 in terms of satisfaction with the procedure (1 = I am not satisfied with the procedure, 10 = I am very satisfied with the procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Zübeyde Özdemir, Study Chair — ethics committee chairman
Locations (2):
- Turkey (Türkiye) (2):
  - Aylin Ceren Şanlı, Istanbul
  - Aylin Ceren, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided
yes